CLINICAL TRIAL: NCT02514668
Title: An Open-label, Dose-escalation and Multi-center Study to Evaluate the Safety, Pharmacokinetics and Efficacy of SAR650984 (Isatuximab) in Patients With Relapsed/Refractory Multiple Myeloma
Brief Title: A Study to Evaluate the Safety, Pharmacokinetics, and Efficacy of Isatuximab in Patients With Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TED14154; U1111-1163-1073 (Other: UTN)
Record Dates: First submitted 2015-07-31; First posted 2015-08-04 (Estimated); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Plasma Cell Myeloma
Keywords: Anti-CD38 monoclonal antibody
MeSH Terms: conditions — Multiple Myeloma | interventions — isatuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Isatuximab (Experimental): Isatuximab (escalating dose) on Days 1, 8, 15, and 22, then Days 1 and 15 in 28-day cycles up to disease progression
  Interventions: Drug: Isatuximab

INTERVENTIONS:
Drug: Isatuximab — Pharmaceutical form: solution for infusion
  Route of administration: intravenous
  Other Names: SAR650984; Sarclisa

SUMMARY:
Primary Objective:

* Part A: To evaluate the safety of SAR650984 (isatuximab) in patients with relapsed/refractory multiple myeloma (RRMM).
* Part B: To evaluate the activity of SAR650984 (isatuximab) as assessed by overall response rate (ORR) in RRMM patients previously treated with daratumumab.

Secondary Objectives:

* Part A:
* To determine the pharmacokinetics (PK) of SAR650984 (isatuximab) in patients with RRMM.
* Part B:
* To evaluate the safety of SAR650984 (isatuximab).
* To evaluate the efficacy of SAR650984 (isatuximab) as assessed by duration of response (DOR), clinical benefit rate (CBR) and progression free survival (PFS).
* To assess the pharmacokinetics (PK) of SAR650984 (isatuximab) and daratumumab at baseline.
* To evaluate the immunogenicity of SAR650984 (isatuximab).

DETAILED DESCRIPTION:
Study duration for an individual patient will include a screening period for inclusion of up to 3 weeks, the treatment period and, a follow up period. Treatment with SAR650984 (isatuximab) may continue until disease progression, unacceptable adverse event, or other reason for discontinuation.

After study treatment discontinuation, an end of treatment visit will be done at 30 days to assess safety and PK, and at 30 and 60 days for anti-drug antibody (ADA). If the ADA is positive at Day 60, ADA will be repeated every 30 days until ADA is negative.

Patients with partial remission or better who discontinue treatment for reasons other than progression of disease will be followed monthly until progression or initiation of subsequent therapy, the final analysis cutoff date, whichever comes first.

ELIGIBILITY:
Inclusion criteria:

Part A

* Patients must have a known diagnosis of multiple myeloma (MM) with evidence of measurable disease, as defined below, and have evidence of disease progression based on International Myeloma Working Group (IMWG) criteria:
* Serum M-protein ≥1g/dL, or urine M-protein ≥200 mg/24 hours, OR
* In the absence of measurable M-protein, serum immunoglobulin free light chain ≥10 mg/dL, and abnormal serum immunoglobulin kappa lambda free light chain ratio.
* Patients must have received at least 3 prior lines of therapy for MM and must include treatment with an immunomodulatory drug (IMiD) (for ≥2 cycles or ≥2 months of treatment) and a proteasome inhibitor (for ≥2 cycles or ≥2 months of treatment). Induction therapy and stem cell transplant (± maintenance) will be considered as one regimen within a line, OR
* Patients whose disease is double refractory to an IMiD and a proteasome inhibitor. For patients who have received more than one type of IMiD and proteasome inhibitor, their disease must be refractory to the most recent one.
* Patients must have achieved a minimal response (MR) or better to at least one prior line of therapy.
* Patients must have received an alkylating agent (for ≥2 cycles or ≥2 months of treatment) either alone or in combination with other MM treatments (history of stem cell transplant is acceptable). Treatment with high-dose Melphalan for stem cell transplantation meets this requirement.
* Signed written informed consent and be willing and able to complete all study-related procedures.

Part B

* Patients must have a known diagnosis of multiple myeloma (MM) with evidence of measurable disease, as defined below, and have evidence of disease progression based on International Myeloma Working Group (IMWG) criteria:
* Serum M-protein ≥1g/dL, or urine M-protein ≥200 mg/24 hours, OR
* In the absence of measurable M-protein, serum immunoglobulin free light chain ≥10 mg/dL, and abnormal serum immunoglobulin kappa lambda free light chain ratio.
* Patients must have received at least 3 cycles of daratumumab treatment with at least 6 weeks from the last treatment with daratumumab to the first study treatment OR at least 2 cycles of daratumumab treatment in case another therapy is given between daratumumab and isatuximab with at least 12 weeks from the last treatment with daratumumab to the first study treatment.
* Patients must have achieved MR or better to at least 1 prior line of therapy.
* Signed written informed consent and be willing and able to complete all study-related procedures.

Exclusion criteria:

* Patients <18 years old.
* Eastern Cooperative Oncology Group (ECOG) performance status >2.
* Poor bone marrow reserve.
* Poor organ function.
* Known intolerance/hypersensitivity to IMiDs, dexamethasone, boron or mannitol, sucrose, histidine, or polysorbate 80.
* Any serious active disease (including clinically significant infection that is chronic, recurrent, or active) or comorbid condition, which, in the opinion of the Investigator, could interfere with the safety, the compliance with the study, or with the interpretation of the results.
* Any severe underlying medical conditions including presence of laboratory abnormalities, which could impair the ability to participate in the study or the interpretation of its results.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2021-12-02 (Actual); Study Completion 2021-12-02 (Actual)

PRIMARY OUTCOMES:
Part A: Dose Limiting Toxicities (DLTs) | Up to 4 weeks
Part A: Number of patients with adverse events (AEs) and changes in laboratory tests and vital signs according to the National Cancer Institute - Common Toxicity Criteria (NCI-CTC) version 4.03 grade scaling | Up to 30 days following the last administration of study treatment or up to 12 months for ongoing related AE, ongoing serious AE and new related AE
Part B: Overall Response Rate (ORR) | 4 months

SECONDARY OUTCOMES:
Assessment of PK parameters: partial area under the serum concentration time curve (AUC) | 1 week after first treatment
Assessment of PK parameters: maximum observed concentration (Cmax) | 1 week after first treatment
Part B: Number of patients with AEs and changes in laboratory tests and vital signs according to the National Cancer Institute - Common Toxicity Criteria (NCI-CTC) version 4.03 grade scaling | Up to 30 days following the last administration of study treatment or up to 12 months for ongoing related AE, ongoing serious AE and new related AE
Part B: Duration of Response (DOR) | Up to 12 months from the last patient in
Part B: Clinical Benefit Rate (CBR) | Up to 12 months from the last patient in
Part B: Progression Free Survival (PFS) | Up to 12 months from the last patient in
Part B: Levels of isatuximab antibodies | Up to 12 months from the last patient in

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (18):
- United States (10):
  - Investigational Site Number 840003, Scottsdale, Arizona
  - Investigational Site Number 840004, San Francisco, California
  - Investigational Site Number 840011, Detroit, Michigan
  - Investigational Site Number 840015, St Louis, Missouri
  - Investigational Site Number 840005, Hackensack, New Jersey
  - Investigational Site Number 840010, Durham, North Carolina
  - Investigational Site Number 840013, Canton, Ohio
  - Investigational Site Number 840001, Nashville, Tennessee
  - Investigational Site Number 840002, Salt Lake City, Utah
  - Investigational Site Number 840006, Milwaukee, Wisconsin
- Czechia (2):
  - Investigational Site Number 203002, Brno
  - Investigational Site Number 203001, Prague
- France (6):
  - Investigational Site Number 250008, Créteil
  - Investigational Site Number 250005, Montpellier
  - Investigational Site Number 250002, Nantes
  - Investigational Site Number 250004, Pessac
  - Investigational Site Number 250001, Poitiers
  - Investigational Site Number 250006, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Mikhael J, Belhadj-Merzoug K, Hulin C, Vincent L, Moreau P, Gasparetto C, Pour L, Spicka I, Vij R, Zonder J, Atanackovic D, Gabrail N, Martin TG, Perrot A, Bensfia S, Weng Q, Brillac C, Semiond D, Mace S, Corzo KP, Leleu X. A phase 2 study of isatuximab monotherapy in patients with multiple myeloma who are refractory to daratumumab. Blood Cancer J. 2021 May 12;11(5):89. doi: 10.1038/s41408-021-00478-4. No abstract available. PMID 33980831